CLINICAL TRIAL: NCT00224705
Title: Efficacy and Safety of the Albumin Dialysis MARS® Therapy in Patients With Fulminant and Subfulminant Hepatic Failure
Brief Title: The MARS® Albumin Dialysis System in Patients With Fulminant and Subfulminant Hepatic Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cecile JOURDAIN, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P030423
Record Dates: First submitted 2005-09-19; First posted 2005-09-23 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2007-07

CONDITIONS: Hepatitis
Keywords: Albumin dialysis; MARS system; Extracorporeal artificial liver support; Fulminant hepatitis; Subfulminant hepatitis; Acute liver failure
MeSH Terms: conditions — Hepatitis; Massive Hepatic Necrosis; Liver Failure, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Molecular Adsorbent Recirculating System (MARS®)

SUMMARY:
The purpose of this study is to improve the survival rate of those patients with acute fulminant hepatitis through treatment with the MARS® extra-corporal liver-purification system by:

1. Reducing the number of patients who die before a graft is available
2. Increasing the chances of survival without a liver transplant
3. Reducing the pre- and post-operative mortality in transplant patients

DETAILED DESCRIPTION:
Patients with fulminant or subfulminant hepatitis with either an indication or a relative contraindication to a liver transplantation, are randomized to two groups:

1. A group treated with the conventional medical intensive treatment (including the hemodialysis techniques, continuous veno-venous hemofiltration or hemodiafiltration, if necessary) and the gold standard surgical treatment (liver transplantation) compared to
2. A group receiving, in addition to the conventional medical intensive treatment, albumin dialysis using the MARS device and the gold standard surgical treatment (liver transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe or sub-severe hepatitis, with an indication or a contraindication to liver transplantation

Exclusion Criteria:

* Sepsis severe not controlled
* Haemorrhage activates not controlled
* Clinical Obviousness of disseminated intravascular coagulation
* Severe Pathology cardiopulmonary (NYHA > or = 2)
* Pregnancy, breast feeding
* Average blood Pressure < 40 mmHg more than 10 minutes in spite of a support by the inotrope
* Nonhepatic coma of origin
* Cholestases extra-hepatitic
* Antecedents of heavy surgery in the 4 previous weeks or surgical problems unsolved
* Absolute counter-indication with hepatic transplantation (extra Neoplasia hepatic evolutionary, irreversible cerebral Attack, irreversible multi-visceral Failure, visceral tares contra-indicating the transplantation)
* Positive serology HIV
* Hepatic Demonstrations of the malignant hemopathies
* Participation in another therapeutic test in the 4 previous weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Patient survival at six months | 6 months

SECONDARY OUTCOMES:
Patient survival at six months without neurological sequelae | 6 months
Patient survival at 1 year | during one year
Graft survival at six months and 1 year | at 6 months and at one year
Number of patients who improve their liver function and no longer need a transplant in each stage of the trial | during one year
Hospital mortality before the transplant | during one year
Evaluation, at different stages, of the progression of the neurological condition (clinical and electroencephalographic stages, Glasgow scale) | during one year
Evaluation at different stages, of the progression of biological parameters, which reflect liver and kidney function | during one year
Evaluation of the safety parameters of the MARS® system (thromboembolism, risk of haemorrhage and infections) | during one year
Economic elements: duration of stay in the Intensive Care Unit (ICU) up to the transplant and after the transplant | during one year
duration of hospitalisation | during one year

CONTACTS AND LOCATIONS:
Overall Officials: Faouzi SALIBA, Pr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Paul Brousse, Villejuif, France

REFERENCES:
- [Background] Novelli G, Rossi M, Pretagostini R, Novelli L, Poli L, Ferretti G, Iappelli M, Berloco P, Cortesini R. A 3-year experience with Molecular Adsorbent Recirculating System (MARS): our results on 63 patients with hepatic failure and color Doppler US evaluation of cerebral perfusion. Liver Int. 2003;23 Suppl 3:10-5. doi: 10.1034/j.1478-3231.23.s.3.4.x. PMID 12950955
- [Derived] Saliba F, Camus C, Durand F, Mathurin P, Letierce A, Delafosse B, Barange K, Perrigault PF, Belnard M, Ichai P, Samuel D. Albumin dialysis with a noncell artificial liver support device in patients with acute liver failure: a randomized, controlled trial. Ann Intern Med. 2013 Oct 15;159(8):522-31. doi: 10.7326/0003-4819-159-8-201310150-00005. PMID 24126646